CLINICAL TRIAL: NCT03648008
Title: Postoperative Analgesic Effect of Hydromorphone on Chinese Patients Receiving Partial Pulmonary Resection Under Video-assisted Thoracoscopy
Brief Title: Postoperative Analgesic Effect of Hydromorphone on Partial Pulmonary Resection Under Video-assisted Thoracoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-014
Record Dates: First submitted 2018-08-13; First posted 2018-08-27 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Pain, Postoperative; Thoracic Surgery, Video-Assisted
MeSH Terms: conditions — Pain, Postoperative | interventions — Hydromorphone; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group M (Active Comparator): Drug: Morphine Background: No Bolus infusion: 0.015 mg*kg-1
  Interventions: Drug: Morphine
- Group NBH (Experimental): Drug: Hydromorphone Background: No Bolus infusion: 0.002 mg*kg-1
  Interventions: Drug: Hydromorphone
- Group BH (Experimental): Drug: Hydromorphone Background: 0.002 mg*kg-1*h-1 Bolus infusion: 0.002 mg*kg-1
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Hydromorphone — 0.002 mg*kg-1 bolus with 0.002 mg*kg-1 background infusion for group BH 0.002 mg*kg-1 bolus without background infusion for group NBH Drug is administered through PCIA pump.
  Arms: Group BH; Group NBH
Drug: Morphine — 0.015 mg*kg-1 bolus without background infusion for group M Drug is administered through PCIA pump.
  Arms: Group M

SUMMARY:
Postoperative pain remains relatively high within 48h for Chinese patients who receive video-assisted thoracoscopic surgery. Multimodal analgesia combines several agents and/or techniques to function on diverse nociceptive mechanisms to enhance pain relief and lessen side effect. Hydromorphone is a hydrogenated ketone of morphine and approximately 5-10 times more potent. There lacks about efficacy and efficiency of hydromorphone in electrical pump for patient controlled intravenous analgesic (PCIA).

ELIGIBILITY:
Inclusion Criteria:

* 70≥ Age ≥18
* Selective operation lung section with video-assisted thoracic surgery (VATS)
* III ≥ American Society of Anesthesiologists classification (ASA classification) ≥I
* Patients informed and agreed to join the study

Exclusion Criteria:

* Abnormal function of liver and kidney
* Allergic- dependence history of alcohol, opioids and Local anesthetics
* No noncompliance
* Mental disease history，language communication disorder，cicatricial diathesis
* Underweight or overweight（BMI<18 or >30)
* Patients not suitable for clinical subjects for other reasons
* Sedatives, analgesics, antiemetic drugs and anti pruritus drugs were used within 24 hours before the operation.
* History of previous abnormal anaesthesia
* Women during pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Rest pain assessment at 0.5 hour after tracheal extubation | 0.5 hour after tracheal extubation
  Visual Analogue Scale/Score to assess pain at rest. VAS range from 0 to 100 millimeter. And 0 stands for no pain, while 100 stands for worst pain. Lower value is better.
Rest pain assessment at 8 p.m. surgery day | 8 p.m. at surgery day
  Visual Analogue Scale/Score to assess pain at rest. VAS range from 0 to 100 millimeter. And 0 stands for no pain, while 100 stands for worst pain. Lower value is better.
Activity pain assessment at 8 p.m. surgery day | 8 p.m. at surgery day
  Visual Analogue Scale/Score to assess pain on coughing. VAS range from 0 to 100 millimeter. And 0 stands for no pain, while 100 stands for worst pain. Lower value is better.
Rest pain assessment at 8 a.m. at first day after surgery | 8 a.m. at first day after surgery
  Visual Analogue Scale/Score to assess pain at rest. VAS range from 0 to 100 millimeter. And 0 stands for no pain, while 100 stands for worst pain. Lower value is better.
Activity pain assessment at 8 a.m. at first day after surgery | 8 a.m. at first day after surgery
  Visual Analogue Scale/Score to assess pain on coughing. VAS range from 0 to 100 millimeter. And 0 stands for no pain, while 100 stands for worst pain. Lower value is better.
Rest pain assessment at 8 p.m. at first day after surgery | 8 p.m. at first day after surgery
  Visual Analogue Scale/Score to assess pain at rest. VAS range from 0 to 100 millimeter. And 0 stands for no pain, while 100 stands for worst pain. Lower value is better.
Activity pain assessment at 8 p.m. at first day after surgery | 8 p.m. at first day after surgery
  Visual Analogue Scale/Score to assess pain on coughing. VAS range from 0 to 100 millimeter. And 0 stands for no pain, while 100 stands for worst pain. Lower value is better.
Rest pain assessment at 8 a.m. at second day after surgery | 8 a.m. at second day after surgery
  Visual Analogue Scale/Score to assess pain at rest. VAS range from 0 to 100 millimeter. And 0 stands for no pain, while 100 stands for worst pain. Lower value is better.
Activity pain assessment at 8 a.m. at second day after surgery | 8 a.m. at second day after surgery
  Visual Analogue Scale/Score to assess pain on coughing. VAS range from 0 to 100 millimeter. And 0 stands for no pain, while 100 stands for worst pain. Lower value is better.
Rest pain assessment at 8 p.m. at second day after surgery | 8 p.m. at second day after surgery
  Visual Analogue Scale/Score to assess pain at rest. VAS range from 0 to 100 millimeter. And 0 stands for no pain, while 100 stands for worst pain. Lower value is better.
Activity pain assessment at 8 p.m. at second day after surgery | 8 p.m. at second day after surgery
  Visual Analogue Scale/Score to assess pain on coughing. VAS range from 0 to 100 millimeter. And 0 stands for no pain, while 100 stands for worst pain. Lower value is better.
Rest pain assessment at 8 a.m. at third day after surgery | 8 a.m. at third day after surgery
  Visual Analogue Scale/Score to assess pain at rest. VAS range from 0 to 100 millimeter. And 0 stands for no pain, while 100 stands for worst pain. Lower value is better.
Activity pain assessment at 8 a.m. at third day after surgery | 8 a.m. at third day after surgery
  Visual Analogue Scale/Score to assess pain on coughing. VAS range from 0 to 100 millimeter. And 0 stands for no pain, while 100 stands for worst pain. Lower value is better.
Rest pain assessment at 8 p.m. at third day after surgery | 8 p.m. at third day after surgery
  Visual Analogue Scale/Score to assess pain at rest. VAS range from 0 to 100 millimeter. And 0 stands for no pain, while 100 stands for worst pain. Lower value is better.
Activity pain assessment at 8 p.m. at third day after surgery | 8 p.m. at third day after surgery
  Visual Analogue Scale/Score to assess pain on coughing. VAS range from 0 to 100 millimeter. And 0 stands for no pain, while 100 stands for worst pain. Lower value is better.

SECONDARY OUTCOMES:
Ratio of Nausea | 8 p.m. at surgery day
  Record whether patients experience nausea
Ratio of Vomiting | 8 p.m. at surgery day
  Record whether patients experience vomiting and how many times do they experience
Ratio of Nausea | 8 a.m. at first day after surgery
  Record whether patients experience nausea
Ratio of Vomiting | 8 a.m. at first day after surgery
  Record whether patients experience vomiting and how many times do they experience
Ratio of Nausea | 8 p.m. at first day after surgery
  Record whether patients experience nausea
Ratio of Vomiting | 8 p.m. at first day after surgery
  Record whether patients experience vomiting and how many times do they experience
Ratio of Nausea | 8 a.m. at second day after surgery
  Record whether patients experience nausea
Ratio of Vomiting | 8 a.m. at second day after surgery
  Record whether patients experience vomiting and how many times do they experience
Ratio of Nausea | 8 p.m. at second day after surgery
  Record whether patients experience nausea
Ratio of Vomiting | 8 p.m. at second day after surgery
  Record whether patients experience vomiting and how many times do they experience
Ratio of Nausea | 8 a.m. at third day after surgery
  Record whether patients experience nausea
Ratio of Vomiting | 8 a.m. at third day after surgery
  Record whether patients experience vomiting and how many times do they experience
Ratio of Nausea | 8 p.m. at third day after surgery
  Record whether patients experience nausea
Ratio of Vomiting | 8 p.m. at third day after surgery
  Record whether patients experience vomiting and how many times do they experience
Total Analgesia usage | 8 p.m. at surgery day
  Sum up any extra analgesia when analgesic failure (VAS persistently > 4) with PCIA pump
Total Antiemetic usage | 8 p.m. at surgery day
  Sum up any antiemetic
Total Analgesia usage | 8 a.m. at first day after surgery
  Sum up any extra analgesia when analgesic failure (VAS persistently > 4) with PCIA pump from last time point
Total Antiemetic usage | 8 p.m. at first day after surgery
  Sum up any antiemetic from last time point
Total Analgesia usage | 8 p.m. at first day after surgery
  Sum up any extra analgesia when analgesic failure (VAS persistently > 4) with PCIA pump from last time point
Total Analgesia usage | 8 a.m. at second day after surgery
  Sum up any extra analgesia when analgesic failure (VAS persistently > 4) with PCIA pump from last time point
Total Antiemetic usage | 8 a.m. at second day after surgery
  Sum up any antiemetic from last time point
Total Analgesia usage | 8 p.m. at second day after surgery
  Sum up any extra analgesia when analgesic failure (VAS persistently > 4) with PCIA pump from last time point
Total Antiemetic usage | 8 p.m. at second day after surgery
  Sum up any antiemetic from last time point
Total Analgesia usage | 8 a.m. at third day after surgery
  Sum up any extra analgesia when analgesic failure (VAS persistently > 4) with PCIA pump from last time point
Total Antiemetic usage | 8 a.m. at third day after surgery
  Sum up any antiemetic from last time point
Total Analgesia usage | 8 p.m. at third day after surgery
  Sum up any extra analgesia when analgesic failure (VAS persistently > 4) with PCIA pump from last time point
Total Antiemetic usage | 8 p.m. at third day after surgery
  Sum up any antiemetic from last time point

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Doctor, Study Chair — Zhejiang University
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No